CLINICAL TRIAL: NCT04029142
Title: Screening for Hemoglobinopathies in Pregnant Women
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01065; sp19Amstad
Record Dates: First submitted 2019-07-17; First posted 2019-07-23 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Hemoglobinopathies
Keywords: thalassemia; sickle cell anaemia; molecular genetic analysis
MeSH Terms: conditions — Hemoglobinopathies; Thalassemia; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Review of routine lab data — Review of routine lab data from pregnant women (first trimester)

SUMMARY:
This prospective monocentric study project is to identify hemoglobinopathies in pregnant women in order to optimize antenatal care and to investigate the prevalence of hemoglobinopathies in pregnant women in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women seen at the Frauenklinik at University Hospital Basel

Exclusion Criteria:

* pregnant women with already known hemoglobinopathy
* refusal of participation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women seen at the Frauenklinik at University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 1785 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
identification of hemoglobinopathies | single time point assessment at baseline
  identification of hemoglobinopathies by investigating routine lab samples

CONTACTS AND LOCATIONS:
Overall Officials: Irene Hoesli, Prof. Dr., Principal Investigator — Frauenklinik Universitätsspital Basel
Locations (1):
- Frauenklinik University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Amstad Bencaiova G, Geissler F, Hoesli I. Cohort profile: targeted antenatal screening for haemoglobinopathies in Basel. BMJ Open. 2020 Jul 22;10(7):e035735. doi: 10.1136/bmjopen-2019-035735. PMID 32699163